CLINICAL TRIAL: NCT00426517
Title: Allogeneic and Matched Unrelated Donor Stem Cell Transplantation for Congenital Immunodeficiencies or Patients With Autoinflammatory/Immunodysregulatory Conditions: Busulfan-Based Conditioning With Campath- 1H or h-ATG, Radiation, and Sirolimus
Brief Title: Donor Stem Cell Transplantation for Congenital Immunodeficiencies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 070075; 07-I-0075 (Other: NIHCC)
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2019-11-01

CONDITIONS: Inherited Immune Deficiencies
Keywords: MUD Transplant; Transplant; AlloPBSC; HLA Matched Transplant; BMT; Congenital Immunodeficiency; Bone Marrow Transplant
MeSH Terms: interventions — Alemtuzumab; Busulfan; Dosage Forms; Whole-Body Irradiation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Matched related donor stem cell transplant (Experimental): Conditioning with Campath 1 mg/kg total dose given intravenously over 5 days, Busulfan 10 mg/kg total dose given intravenously over 2 days
  Interventions: Drug: Campath 1H; Drug: Busulfan; Drug: Sirolimus or equivalent based on response
- Matched unrelated donor stem cell transplant (Experimental): Conditioning with Campath 1 mg/kg total dose given intravenously over 5 days, Busulfan 5 mg/kg total dose given intravenously over 2 days, and Total Body Irradiation (TBI) 200 cGy in two fractions on the same day
  Interventions: Drug: Campath 1H; Drug: Busulfan; Drug: Total Body Irradiation (TBI); Drug: Sirolimus or equivalent based on response
- Matched unrelated donor stem cell transplant (MUD-non CGD) (Experimental): Conditioning with ATG 40 mg/kg total dose over 4 days IV, Busulfan 5 mg/kg total dose over 2 days IV, and TBI 300 cGy in two fractions at day -2
  Interventions: Drug: Busulfan; Drug: Horse Anti-human Thymocyte Globulin (h-ATG); Drug: Total Body Irradiation (TBI); Drug: Sirolimus or equivalent based on response
- Matched unrelated donor transplant (MUD-CGD) cord blood (Experimental): Conditioning with Campath 1 mg/kg total dose given intravenously over 5 days, Busulfan 5 mg/kg total dose given intravenously over 2 days, and Total Body Irradiation (TBI) 200 cGy in two fractions on the same day
  Interventions: Drug: Campath 1H; Drug: Busulfan; Drug: Total Body Irradiation (TBI); Drug: Sirolimus or equivalent based on response

INTERVENTIONS:
Drug: Campath 1H — Conditioning with Campath 1 mg/kg total dose given intravenously over 5 days
  Other Names: alemtuzumab
  Arms: Matched related donor stem cell transplant; Matched unrelated donor stem cell transplant; Matched unrelated donor transplant (MUD-CGD) cord blood
Drug: Busulfan — Busulfan 5-10 mg/kg total dose given intravenously over 2 days based on patient underlining immune deficiency disorder
  Other Names: Busulfex® (IV formulation)
Drug: Horse Anti-human Thymocyte Globulin (h-ATG) — Conditioning with h-ATG 40 mg/kg total dose over 4 days given intravenously
  Other Names: ATG
  Arms: Matched unrelated donor stem cell transplant (MUD-non CGD)
Drug: Total Body Irradiation (TBI) — TBI 200 - 300 centigray (cGy) in two fractions at day -2 or same day depending on patient underlining immune deficiency disorder
  Other Names: TBI
  Arms: Matched unrelated donor stem cell transplant; Matched unrelated donor stem cell transplant (MUD-non CGD); Matched unrelated donor transplant (MUD-CGD) cord blood
Drug: Sirolimus or equivalent based on response — post Transplantation immunosuppressants
  Other Names: Rapamune®/rapamycin

SUMMARY:
This study uses transplantation to treat patients with problems in their immune system. The immune system cells come from the bone marrow where they grow from special cells called stem cells. Giving patients stem cells from someone else may help to cure many patients with certain immune diseases. This is called 'bone marrow transplantation'. This procedure can have side effects that are life-threatening. To try to make transplantation safer we are using lower doses of the medications used in preparing the patient for the transplant.

'Conditioning' treatments are given to patients to create space in their bone marrow. This lets the cells of the donor go into the bone marrow and produce normal immune cells. This study will use lower doses of a drug called busulfan and lower doses of radiation than what are currently being used in other kinds of bone marrow transplantation for other diseases.

Another problem that can occur with bone marrow transplantation is 'graft-versus-host disease'. This happens when the cells of the donor attacks different parts of the patient s body. This study will use a medicine called sirolimus instead of the usual medicine, cyclosporine, to prevent graft-versus-host disease.

To go onto this study, you must have:

1. A severe immune deficiency, such as chronic granulomatous disease or leukocyte adhesion deficiency.
2. Have problems from the disease that call for stem cell transplantation.
3. You must also be between the ages of 2 and 40 years.

Two groups of patients are included in this study:

1. Patients who have a brother or sister that have stem cells that match the patient. This is known as an allogeneic matched sibling transplant.
2. Patients who do not have a matched sibling donor but have a donor that matches in the National Marrow Donor Program. This is know as matched unrelated donor transplantation.

Patients will have the following procedures:

* To create space in the bone marrow, patients are given two drugs, Campath-1H and busulfan. To prevent the body from getting rid of the donated cells, patients are given sirolimus. On the day before the BMT, patients in the matched unrelated donor group also receive a low-dose of whole-body radiation. This will further improve the chances that the patients body will accept the donor cells.
* Patients will get the donor stem cells through an intravenous (IV) line that goes into a vein in their body. The cells make their way to the bone marrow space and slowly refill the marrow over the next several weeks. Patients will usually stay in the hospital for 30 days after the transplant.
* For the first 3 months after the transplant, patients are watched closely. The patients will have frequent visits to the clinic. During these visits the patient will have a physical examination and blood tests. The doctor and nurse will also check any symptoms the patient may have. At day 100 after the transplant a sample of bone marrow is taken.
* Patients will continue to be followed periodically for at least 5 years after the transplant.

DETAILED DESCRIPTION:
This is an open-label pilot study of HLA-matched allogenic and matched unrelated donor (MUD) hematopoietic stem cell (HSC) transplant (also referred to as peripheral blood stem cell (PBSC) or bone marrow transplant (BMT)) for patients with X-linked severe combined immune deficiency (XSCID). XSCID is caused by mutations in the IL2RG gene encoding the interleukin receptor signaling gamma chain [gamma c]). The study population are older children (greater than or equal to 2 years of age) and adults (less than or equal to 40 years of age) who are experiencing deteriorating and/or dysfunctional immunity and any of a constellation of severe or chronic medical problems warranting transplantation. The study is designed to evaluate whether the use of uniquely designed transplant conditioning and graft-versus-host disease (GvHD) prevention regimens achieve sufficient engraftment of donor hematopoietic stem cells (HSCs) to facilitate robust restoration of cellular immunity (T cell/NK cell number and function) including thymic function, and humoral immunity (B cell number and function) while at the same time enhancing tolerance of the donor graft in a fashion that reduces the occurrence of GvHD but not at significantly enhancing the risk of post-transplant virus infection. One target population are XSCID patients who received matched sibling or haploidentical lymphocyte-depleted transplants as infants with little or no myeloid conditioning, resulting in variable restoration of T cell immunity, but little or no restoration of NK or B cell immunity. Another target population are XSCID patients with partial production or function of gamma c or XSCID patients with clonal somatic reversion of the mutation in the IL2RG gene, who have less severe immune deficiency in childhood. A subset of patients from all of these target XSCID populations may experience progressive deterioration of immune function leading to acute and chronic medical problems that warrant consideration of allogeneic or MUD transplant to restore immunity.

The conditioning and GvHD prevention regimens for this HSC transplant protocol are designed to use mobilized peripheral blood stem cells (PBSC) or bone marrow (BM) (if mobilization is not possible) from either an HLA-matched related sibling donor (alloPBSC) as first choice or from an HLA matched unrelated donor (MUD) for those without an appropriate HLA-matched related sibling donor. If there is no appropriately matched sibling donor nor MUD adult donor available, then an appropriately matched cord blood from the cord blood registries may be used for small children XSCID recipients. For the alloPBSC (or alloBM) transplantation (referred to as Group 1), we propose using a busulfan-based, nonmyeloablative conditioning regimen combined with horse Anti-human Thymocyte Globulin (h-ATG) immune suppression conditioning plus post-transplant sirolimus for tolerance inducing immunosuppressant to prevent GvHD. For the MUD or unrelated cord blood transplantation (referred to as Group 2), we will use a similar conditioning regimen, with a few modifications that include addition of total body irradiation with shielding and reduction in busulfan dosing, changes designed to address the increased risk of graft rejection with HLA-matched but unrelated donor HSC.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS (RECIPIENT)

* Must have confirmed genetic diagnosis of XSCID (common gamma chain disorder) by identification of a mutation in the IL2RG gene or by demonstrating failure to detect gamma c protein in patient immune blood cells.
* Must have sufficient complications from underlying disease to warrant undergoing transplantation as defined as follows:.

Clinical Criteria: (greater than or equal to 1 must be present)

i. Infections (not including molluscum, warts or mucocutaneous candidiasis; see vii and viii below): 3 significant new or chronic active infections during the 2 years preceding evaluation for enrollment, with each infection accounting for one criteria.

Infections are defined as an objective sign of infection (fever >38.30C [1010F] or neutrophilia or pain/redness/swelling or radiologic/ultrasound imaging evidence or typical lesion or histology or new severe diarrhea or cough with sputum production). In addition to one or more of these signs/symptoms of possible infection, there also must be at least 1 of the following criteria as evidence of the attending physician's intent to treat a significant infection (a. and b.) or objective evidence for a specific pathogen causing the infection (c.)

1. Treatment (not prophylaxis) with systemic antibacterial, antifungal or antiviral antibiotics . 14 days OR
2. Hospitalization of any duration for infection OR
3. Isolation of a bacteria, fungus, or virus from biopsy, skin lesion, blood, nasal washing, bronchoscopy, cerebrospinal fluid or stool likely to be an etiologic agent of infection

ii. Chronic pulmonary disease as defined by:

1. Bronchiectasis by x-ray computerized tomography OR
2. Pulmonary function test (PFT) evidence for restrictive or obstructive disease that is . 60% of Predicted for Age OR
3. Pulse oximetry . 94% in room air (if patient is too young to comply with performance of PFTs).

iii. Gastrointestinal enteropathy:

1. Diarrhea-watery stools . 3 times per day (of at least 3 months duration that is not a result of infection as defined in criterion # i. above) OR
2. Endoscopic evidence (gross and histologic) for enteropathy (endoscopy will only be performed if medically indicated) OR
3. Other evidence of enteropathy or bacterial overgrowth syndrome: including malabsorption of fat soluble vitamin(s), abnormal D-xylose absorption, abnormal hydrogen breath test, evidence of protein losing enteropathy (for example increasingly high or frequent dosing of intravenous gamma globulin supplement required to maintain blood IgG level).

iv. Poor nutrition: Requires G-tube or intravenous feeding supplement to maintain weight or nutrition.

v. Auto- or allo-immunity: Examples must include objective physical findings that include, but are not limited to any one of alopecia, severe rashes, uveitis, joint pain with redness or swelling or limitation of movement that is not a result of infection, lupus-like lesions, and granulomas (Does not include auto- or allo-immune enteropathy which is criterion iii). Where possible and appropriate, diagnosis will be supported by histopathology or other diagnostic modality.

vi. Failure to grow in height: . 3rd percentile for age

vii. Skin molluscum contagiosum OR warts (this criterion is satisfied if molluscum consists of 10 lesions or there are two or more lesions at each of two or more widely separated anatomic sites; or there are 3 warts at different anatomic sites at the same time; or the patient has both

molluscum and warts)

viii. Mucocutaneous candidiasis (chronic oral thrush or candida esophagitis or candida intertriginous infection or candida nail infections; must be culture positive to satisfy this criterion)

ix. Hypogammaglobulinemia: requires regular IgG supplementation

Ages 2 years 40 years.

HLA-matched family donor available or an HLA matched unrelated PBSC graft (10/10 or 9/10 mismatch) available, or a minimum of 4/6 HLA matched cord blood product. (If the size of the cord blood graft is less than 3.0 x 10(7) cells, a second appropriate 4/6 or greater match cord blood product must be available).

Must be HIV negative.

Must be able to stay within one hour s travel of the NIH for the first 3 months after transplantation and have a family member or other designated companion to stay with during the post transplant period.

Must provide a durable power of attorney for health care decisions to an appropriate adult relative or guardian in accordance to NIH -200 NIH Durable Power of Attorney for Health Care Decision Making.

If of child-bearing potential, must agree to consistently use contraception throughout study participation and for 3 months post-study. Acceptable forms of contraception are:

* Condoms, male or female, with or without a spermicide
* Diaphragm or cervical cap with spermicide
* Intrauterine device
* Contraceptive pills or patch, Norplant, Depo-Provera, or other FDA-approved contraceptive method
* Male partner has previously undergone a vasectomy

EXCLUSION CRITERIA:

PATIENT (RECIPIENT)

* Eastern Cooperative Oncology Group (ECOG) or equivalent performance status of 3 or more (See Supportive Care guidelines, available at http://intranettst2.cc.nih.gov/bmt/clinicalcare).
* Left ventricular ejection fraction less than 40%.
* Transaminases greater than 5 times upper limit of normal based on the patient s clinical situation and at the discretion of the investigator.
* Liver alkaline phosphatase >10x upper limit of normal based on the patient's clinical situation and at the discretion of the investigator
* Psychiatric disorder or mental deficiency severe enough as to make compliance with the BMT treatment unlikely, and/or making informed consent impossible.
* Major anticipated illness or organ failure incompatible with survival from AlloPBSC, MUD or unrelated cord blood transplant
* Pregnant or lactating.
* HIV positive.
* Uncontrolled seizure disorder.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01-19; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grunebaum E, Mazzolari E, Porta F, Dallera D, Atkinson A, Reid B, Notarangelo LD, Roifman CM. Bone marrow transplantation for severe combined immune deficiency. JAMA. 2006 Feb 1;295(5):508-18. doi: 10.1001/jama.295.5.508. PMID 16449616
- [Background] Winkelstein JA, Marino MC, Johnston RB Jr, Boyle J, Curnutte J, Gallin JI, Malech HL, Holland SM, Ochs H, Quie P, Buckley RH, Foster CB, Chanock SJ, Dickler H. Chronic granulomatous disease. Report on a national registry of 368 patients. Medicine (Baltimore). 2000 May;79(3):155-69. doi: 10.1097/00005792-200005000-00003. PMID 10844935
- [Background] Johnston RB Jr. Clinical aspects of chronic granulomatous disease. Curr Opin Hematol. 2001 Jan;8(1):17-22. doi: 10.1097/00062752-200101000-00004. PMID 11138621
- [Background] Roesler J, Brenner S, Bukovsky AA, Whiting-Theobald N, Dull T, Kelly M, Civin CI, Malech HL. Third-generation, self-inactivating gp91(phox) lentivector corrects the oxidase defect in NOD/SCID mouse-repopulating peripheral blood-mobilized CD34+ cells from patients with X-linked chronic granulomatous disease. Blood. 2002 Dec 15;100(13):4381-90. doi: 10.1182/blood-2001-12-0165. Epub 2002 Aug 1. PMID 12393624
- [Background] Kang EM, de Witte M, Malech H, Morgan RA, Phang S, Carter C, Leitman SF, Childs R, Barrett AJ, Little R, Tisdale JF. Nonmyeloablative conditioning followed by transplantation of genetically modified HLA-matched peripheral blood progenitor cells for hematologic malignancies in patients with acquired immunodeficiency syndrome. Blood. 2002 Jan 15;99(2):698-701. doi: 10.1182/blood.v99.2.698. PMID 11781257
- [Background] Horwitz ME, Barrett AJ, Brown MR, Carter CS, Childs R, Gallin JI, Holland SM, Linton GF, Miller JA, Leitman SF, Read EJ, Malech HL. Treatment of chronic granulomatous disease with nonmyeloablative conditioning and a T-cell-depleted hematopoietic allograft. N Engl J Med. 2001 Mar 22;344(12):881-8. doi: 10.1056/NEJM200103223441203. PMID 11259721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Started | 7 | 36 | 3 | 2
Completed | 7 | 36 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood | Total
Number analyzed (Participants) | 7 | 36 | 3 | 2 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 23 | 3 | 2 | 31
  Between 18 and 65 years | 4 | 13 | 0 | 0 | 17
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 0 | 5
  Male | 5 | 33 | 3 | 2 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 0 | 1 | 5
  Not Hispanic or Latino | 7 | 32 | 3 | 1 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 5 | 30 | 3 | 0 | 38
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stem Cell Transplant Engraftment
Description: Engraftment of allogeneic or matched unrelated (including cord blood) hematopoietic progenitor cells using moderate-dose busulfan and Campath-1H with or without whole body irradiation so as to attain phenotypic correction of congenital immunodeficiencies.
Time Frame: 1 year
Population: The analyses include only those who underwent transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Participants | 7 | 31 | 3 | 0

2. Secondary Outcome: Engraftment Without Development of GVHD
Description: Participants who achieved engraftment without development of graft versus host disease (GVHD).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Participants | 6 | 30 | 3 | NA — Subjects did not engraft

3. Secondary Outcome: Participants With Established Stable Mixed Chimerism
Description: Number of participants with myeloid chimerism of greater than 10% of donor cells at 1 year post transplant
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Participants | 7 | 30 | 3 | NA — Subjects did not engraft

4. Secondary Outcome: Days to CD3 Count Greater Than 100 u/L
Description: Rapidity of immune reconstitution based on number of days to CD3 count greater than 100 u/L.
Time Frame: 1 year
Population: The analyses include only those who underwent transplant
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Days | 355 (201.8) | 284 (296.64) | 16 (3.46) | NA (NA) — Subjects did not engraft

5. Secondary Outcome: Days to Absolute Neutrophil Recovery (ANC)
Description: Recovery is defined as an absolute neutrophil count (ANC) of ≥ 0.5 x 109 /L (500/mm3 ) for three consecutive laboratory values obtained on different days. Date of ANC recovery is the date of the first of three consecutive laboratory values where the ANC is ≥ 0.5 x 109 /L.
Time Frame: 1 year
Population: The analyses include only those who underwent transplant
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Days | 19.42 (4.57) | 77.44 (192.34) | 25.5 (15.88) | NA (NA) — Subjects did not engraft

6. Secondary Outcome: Number of RBC Transfusions Per Subject
Description: Average number of red blood cell (RBC) transfusion per subject
Time Frame: 1 year
Population: The analyses include only those who underwent transplant
Measure: Mean (Standard Deviation); unit: transfusions per person
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
transfusions per person | 1.71 (1.79) | 7.08 (12.18) | 4 (1) | NA (NA) — Subjects did not engraft

7. Secondary Outcome: Days to Platelet Recovery
Description: Platelet recovery is defined as platelet value ≥ 20 × 109/L for three consecutive days and no platelet transfusions administered for previous seven consecutive days. The date of platelet recovery is the date of the first of three consecutive laboratory values ≥ 20 × 109/L.
Time Frame: 1 year
Population: The analyses include only those who underwent transplant
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Days | 31 (20.21) | 31.9 (30.48) | 32.6 (20.31) | NA (NA) — Subjects did not engraft

8. Secondary Outcome: Incidence of Cytomegalovirus (CMV) Disease
Description: Number of events of Cytomegalovirus disease based on clinical sequelae that requires treatment (not reactivation)
Time Frame: 1 year
Population: The analyses include only those who underwent transplant
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
Number analyzed (Participants) | 7 | 36 | 3 | 2
Number of events | 0 (0) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Matched Related Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood
All-Cause Mortality (participants affected / at risk) | 0/7 | 9/36 | 1/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/36 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/7 | 17/36 | 1/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matched Related Donor Stem Cell Transplant (N=7) | Matched Unrelated Donor Stem Cell Transplant (N=36) | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) (N=3) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood (N=2)
Evans syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Post transplant lymphoproliferative disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Engraft failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matched Related Donor Stem Cell Transplant (N=7) | Matched Unrelated Donor Stem Cell Transplant (N=36) | Matched Unrelated Donor Stem Cell Transplant (MUD-non CGD) (N=3) | Matched Unrelated Donor Transplant (MUD-CGD) Cord Blood (N=2)
Thyroiditis (Endocrine disorders) | 0 | 2 | 0 | 0
Acute graft versus host disease in intestine (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0
Chronic graft versus host disease in skin (Immune system disorders) | 1 | 2 | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 5 | 0 | 0
Engraft failure (Injury, poisoning and procedural complications) | 0 | 5 | 0 | 2
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Acute graft versus host disease in skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
No limitations. Treatment of a rare disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-12-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT00426517/Prot_SAP_000.pdf